CLINICAL TRIAL: NCT02359617
Title: Continuous Glucose Sensing at the Site of Subcutaneous Insulin Administration: Evaluation of a Novel Single-Port Treatment Approach in Type 1 Diabetic Patients During a 1-Day Stay in a Clinical Research Center and a 6-Day Period at Home
Brief Title: Continuous Glucose Sensing at the Site of Subcutaneous Insulin Administration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Collaborators: European Commission (Other)
Responsible Party: Principal Investigator, Pieber Thomas, MD, MD, Prof. of Medicine, Medical University of Graz
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Single-Port@Home-01
Record Dates: First submitted 2015-01-28; First posted 2015-02-10 (Estimated); Last update posted 2015-04-27 (Estimated); Status verified 2015-04

CONDITIONS: Type 1 Diabetes
Keywords: continuous glucose sensor; subcutaneous insulin infusion; closed-loop glucose control; type 1 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- glucose sensing and insulin delivery (Experimental): Subcutaneous insulin delivery with an insulin pump plus glucose sensing with a continuous glucose sensor placed at the site of subcutaneous insulin delivery.
  In parallel, capillary glucose determinations using a conventional glucose meter as well as glucose sensing in subcutaneous, insulin-unexposed tissue using a continuous glucose sensor.
  Interventions: Drug: insulin delivery; Device: glucose sensing

INTERVENTIONS:
Drug: insulin delivery — Subcutaneous insulin (100 U/ml, NovoRapid®; Novo Nordisk, Bagsvaerd, Denmark) delivery with an insulin pump (Vibe-TM; Animas Corp., West Chester, PA, USA) and an insulin infusion cannula (SOF-SET MICRO QR 6mm; Medtronic MiniMed, USA) placed at the same site as the continuous glucose sensor.
Device: glucose sensing — Glucose sensing with a continuous glucose sensor (Dexcom G4 Platinum Sensor; Dexcom Inc., San Diego, USA) placed at the site of subcutaneous insulin delivery.

SUMMARY:
The study seeks to evaluate a novel treatment approach for performing continuous real-time glucose sensing and insulin delivery at the same subcutaneous tissue site.

DETAILED DESCRIPTION:
The treatment of type 1 diabetes usually comprises the measurement of glucose in blood obtained by finger pricking and the administration of insulin via subcutaneous bolus injection or continuous subcutaneous infusion.

This study seeks to test a new treatment approach where glucose sensing and insulin administration are combined and performed at a single subcutaneous tissue site (single-port treatment approach). A single-port device consisting of a continuous glucose sensor and an insulin infusion cannula is inserted into the subcutaneous tissue of 10 type-1 diabetes patients and used for insulin infusion and simultaneous glucose sensing over a 7-day period. The performance of the single-port device is assessed by comparing the obtained glucose readings with those of a blood glucose meter and an additionally worn control sensor.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 65 years of age, both inclusive
* Type 1 diabetes treated with Continuous Subcutaneous Insulin Infusion (CSII)
* HbA1C < 10%
* Signed informed consent before any study-related activities

Exclusion Criteria:

* Severe acute diseases
* Clinically overt diabetic complications
* Mental incapacity, unwillingness or language barriers precluding adequate understanding or co-operation
* Taking of any vasoactive substances or anticoagulation medication
* Diseases of the skin which could interfere with application of the catheters and Sensors as judged by the investigator
* Pregnancy, breastfeeding, intention of becoming pregnant or not using adequate contraception.
* Increased tendency towards development of hypoglycaemia
* Any disease or condition which the investigator or treating physician feels would interfere with the trial or the safety of the subject
* Concurrent participation in another study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-02; Primary Completion 2014-10 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Mean absolute relative difference between sensor readings and capillary glucose readings | 7 days
  Mean absolute relative differences calculated by determining the mean of the absolute value of the percentage difference between paired sensor and capillary glucose concentration

CONTACTS AND LOCATIONS:
Overall Officials: Thomeas R Pieber, MD, Principal Investigator — Medical University of Graz, Internal Medicine, Endocrinology and Metabolism
Locations (1):
- Medical University of Graz, Graz, Styria, Austria